CLINICAL TRIAL: NCT02546271
Title: A Small-group Intervention to Reduce HIV Sexual Transmission Risk Behavior Among HIV-positive Men Who Have Sex With Men
Acronym: GPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Trevor Hart, Dr. Trevor hart, Toronto Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIHR 194226
Record Dates: First submitted 2015-09-04; First posted 2015-09-10 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Risk Behavior
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): GPS program - an 8-week, peer-led group counselling program using motivational interviewing techniques.
  Interventions: Behavioral: GPS

INTERVENTIONS:
Behavioral: GPS

SUMMARY:
Gay Poz Sex (GPS) is an HIV prevention and sexual health promotion program for HIV-positive gay and bisexual men, which takes place in a group counselling format. All participants provided written informed consent at the outset of the study. Eligible participants filled out a 1-hour computer-assisted self-interview questionnaire. Subsequently, participants attended seven 2-hour group sessions, led by 2 peer facilitators, who were HIV-positive gay men, in groups of 5-8 men. Immediately and 3 months following the completion of the GPS program, participants were scheduled to attend a 1-hour session to complete the same questionnaire package. Participants received an honorarium and a list of community resources, including mental health or substance use counseling services, at the end of each assessment. Participants also participated in a program evaluation interview at the 3-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the study, participants had to:

1. identify as male,
2. report engaging in condomless anal sex with another male during the past 3 months,
3. self-report an HIV-positive status,
4. be over the age of 18 years old, and
5. be able to speak and read in English.

Exclusion Criteria:

* Self-reported female gender,
* no condomless anal sex with another male during past 3 months,
* HIV-negative

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Serodiscordant condomless anal sex with a casual partner | Past 3 months
  Condomless anal sex with an HIV-negative or unknown serostatus casual partner

SECONDARY OUTCOMES:
Seroconcordant condonmless anal sex with a casual partner | Past 3 months
  Condomless anal sex with an HIV-positive casual partner

CONTACTS AND LOCATIONS:
Overall Officials: Trevor A Hart, PhD, Principal Investigator — Toronto Metropolitan University

REFERENCES:
- [Derived] Hart TA, Stratton N, Coleman TA, Wilson HA, Simpson SH, Julien RE, Hoe D, Leahy B, Maxwell J, Adam BD. A Pilot Trial of a Sexual Health Counseling Intervention for HIV-Positive Gay and Bisexual Men Who Report Anal Sex without Condoms. PLoS One. 2016 Apr 7;11(4):e0152762. doi: 10.1371/journal.pone.0152762. eCollection 2016. PMID 27054341